CLINICAL TRIAL: NCT03677401
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Pruritus in Adults With Prurigo Nodularis
Brief Title: Study of the Efficacy, Safety and Tolerability of Serlopitant for the Treatment of Pruritus (Itch) With Prurigo Nodularis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-106; 2017-004210-25 (EudraCT Number)
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Prurigo Nodularis
MeSH Terms: conditions — Pruritus | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg Serlopitant Tablets (Experimental)
  Interventions: Drug: 5mg Serlopitant Tablets
- Matching Placebo Tablets (Placebo Comparator)
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: 5mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737
  Arms: 5 mg Serlopitant Tablets
Drug: Placebo Tablets — Placebo Tablets
  Arms: Matching Placebo Tablets

SUMMARY:
Study of the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with prurigo nodularis

ELIGIBILITY:
Inclusion Criteria (Subjects must meet the following criteria to be randomized into the study:

1. Male or female, age 18 years or older at consent.
2. Prurigo nodularis (PN), with at least ten nodules on at least two different body surface areas.
3. Idiopathic PN, or an identified pruritic condition associated with the PN with persistent pruritus despite at least 6 weeks of optimized and stable treatment of the underlying condition.
4. The worst pruritus is identified as within the areas of the PN lesions, with a Worst-Itch Numeric Rating Scale (WI-NRS) score in the 24-hour period prior to the Screening visit, and average weekly WI-NRS score in each of the 2 weeks prior to Baseline visit indicating an appropriate pruritus level for the study.
5. Female subjects of childbearing potential must be willing to practice highly effective contraception until 5 weeks after last dose of study drug.
6. Willing and able to complete daily eDiary entries within a consistent timeframe for the duration of the study.
7. Willing and able to comply with study visits and study related requirements including providing written informed consent.

Exclusion Criteria (Subjects who meet any of the following criteria are not eligible for participation in the study):

1. Prior treatment with serlopitant.
2. Active pruritic skin disease, other than PN, within 6 months (with the exception of acute dermatoses such as contact dermatitis, sunburn, viral exanthem, which have been resolved for longer than 4 weeks).
3. Treatment with any of the following therapies within 4 weeks.

   1. Other neurokinin-1 receptor antagonists (e.g., aprepitant, fosaprepitant, rolapitant).
   2. Systemic or topical immunosuppressive/immunomodulatory therapies.
   3. Systemic therapies with recognized anti-pruritic properties.
   4. Strong cytochrome-P 3A4 inhibitors.
   5. Use of an indoor tanning facility, or natural sun exposure resulting in significant tanning or sunburn.
4. Treatment with topical anti-pruritic therapies within 2 weeks.
5. Treatment with biologic therapies within 8 weeks or 5 half-lives, whichever is longer.
6. Treatment with any investigational therapy within 4 weeks (8 weeks for investigational biologic therapies) or 5 half-lives, whichever is longer.
7. Serum creatinine, total bilirubin, alanine aminotransferase or aspartate aminotransferase > 2.5 times the upper limit of normal during screening.
8. Untreated or inadequately treated thyroid adrenal, or pituitary nodules or disease, or history of thyroid malignancy.
9. Malignancy within 5 years prior to enrollment (exception for non-melanoma cutaneous malignancies).
10. Relevant major psychiatric diagnosis in the past 3 years, such as major depressive disorder, bipolar disorder, schizophrenia, psychotic disorder, intellectual disability, severe alcohol use disorder.
11. Documented history of parasitic infection, including skin parasites such as scabies, within 8 weeks.
12. Any medical condition or disability that could interfere with the assessment of safety or efficacy in this study or compromise the safety of the subject.
13. History of hypersensitivity to serlopitant or any of its components.
14. Currently pregnant or breastfeeding or planning to become pregnant during the study.
15. Planned or anticipated major surgical procedure or other activity that would interfere with the subject's ability to comply with protocol-mandated assessments during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Stander, MD, Principal Investigator — Universitätsklinikum Münster Klinik für Hautkrankheiten Zentrale Studienkoordination für innovative Dermaologie (ZID); Jacek Szepietowski, MD, Ph.D, Principal Investigator — Lukasz Matusiak 4HEALTH; Franz Josef Legat, MD, Principal Investigator — Medizinische Universität Graz
Locations (40):
- Austria (3):
  - Study Site 649, Graz
  - Study Site 648, Linz
  - Study Site 650, Vienna
- Germany (20):
  - Study Site 623, Bad Bentheim
  - Study Site 607, Berlin
  - Study Site 641, Berlin
  - Study Site 600, Bielefeld
  - Study Site 617, Bochum
  - Study Site 608, Bonn
  - Study Site 642, Buxtehude
  - Study Site 606, Dresden
  - Study Site 621, Erlangen
  - Study Site 602, Frankfurt am Main
  - Study Site 639, Hamburg
  - Study Site 605, Heidelberg
  - Study Site 611, Leipzig
  - Study Site 620, Mahlow
  - Study Site 614, Mainz
  - Study Site 601, Münster
  - Study Site 618, Osnabrück
  - Study Site 640, Potsdam
  - Study Site 615, Selters
  - Study Site 643, Stuttgart
- Poland (17):
  - Study Site 636, Bydgoszcz
  - Study Site 628, Iwonicz-Zdrój
  - Study Site 633, Krakow
  - Study Site 624, Krakow
  - Study Site 635, Krakow
  - Study Site 629, Lodz
  - Study Site 631, Olsztyn
  - Study Site 625, Osielsko
  - Study Site 645, Poznan
  - Study Site 644, Poznan
  - Study Site 634, Rzeszów
  - Study Site 638, Szczecin
  - Study Site 632, Torun
  - Study Site 627, Warsaw
  - Study Site 637, Wroclaw
  - Study Site 630, Wroclaw
  - Study Site 647, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 40 sites in US from 29 August 2018 to 06 February 2020. All psrticipants who met the study entry criteria were randomized in a 1:1 ratio to receive daily oral doses of serlopitant 5 mg or placebo.
Pre-assignment Details: During the screening period (4 weeks), all participants were evaluated for eligibility and chronic pruritic conditions frequently associated with Prurigo Nodularis. Participants were to complete an electronic diary (eDiary) at the Screening visit.
Groups:
- Placebo: Randomized participants received daily oral doses of placebo following an initial 3-tablet loading dose on Day 1. Starting on Day 2, participants took 1 tablet per day until the completion of the 10-week treatment period.
- Serlopitant 5 mg: Randomized participants received daily oral doses of serlopitant 5 mg following an initial 3-tablet loading dose on Day 1. Starting on Day 2, participants took 1 tablet per day until the completion of the 10-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Serlopitant 5 mg
Started | 148 | 147
Completed | 138 | 129
Not Completed | 10 | 18
Not completed — Adverse Event | 4 | 14
Not completed — Lack of Efficacy | 3 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Sponsor decision | 0 | 1
Not completed — Reason Unspecified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Serlopitant 5 mg | Total
Number analyzed (Participants) | 148 | 147 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.97) | 57.5 (15.33) | 58.0 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 98 | 192
  Male | 54 | 49 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 145 | 145 | 290
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Worst Itch Numeric Rating Scale (WI-NRS) 4-point Responder Rate at Week 10
Description: During the study, WI-NRS assessments were reported by the participant via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self reported, instrument for measurement of itch intensity and participants were asked to rate the intensity of their itch on an 11- point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity. A participant was a 4-point responder if their change from baseline is ≤ -4 (i.e. a decrease of at least 4).
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Percentage of participants
  Success | 18.95 | 25.90
  Failure | 81.05 | 74.10
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority — P-value from a Cochran-Mantel- Haenszel (CMH) test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation; p = 0.158, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percent of Participants With WI-NRS 4-point Responder Rate at Week 4
Description: as for outcome 1
Time Frame: At Week 4
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
percentage of participants
  Success | 11.49 | 12.63
  Failure | 88.51 | 87.37
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority — P-value from a CMH test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation; p = 0.750, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent of Participants With WI-NRS 4-point Responder Rate at Week 2
Description: as for outcome 1
Time Frame: At Week 2
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
percentage of participants
  Success | 6.76 | 5.55
  Failure | 93.24 | 94.45
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.674, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change From Baseline in WI-NRS at Weeks 2, 4, 6, and 10
Description: During the study, WI-NRS assessments were reported by the participant via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self reported, instrument for measurement of itch intensity and participants were asked to rate the intensity of their itch on an 11- point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity.
Time Frame: At Weeks 2, 4, 6, and 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Score on a scale
  Change from Baseline at Week 2 | -0.94 (1.470) | -1.25 (1.496)
  Change from Baseline at Week 4 | -1.42 (1.908) | -1.60 (1.955)
  Change from Baseline at Week 6 | -1.61 (2.105) | -1.93 (2.182)
  Change from Baseline at Week 10 | -1.86 (2.334) | -2.24 (2.543)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority — P-values, least squares means (LS Mean) and standard deviations (LS SD) from an analysis of covariance (ANCOVA) with treatment group and stratification factor as fixed effects, and baseline value as a covariate; p = 0.060, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.401, ANCOVA — P-values, LS Mean and LS SD from ANCOVA with treatment group and stratification factor as fixed effects, and baseline value as a covariate
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 6; Test type: Superiority — P-values, LS Mean and LS SD from ANCOVA with treatment group and stratification factor as fixed effects, and baseline value as a covariate; p = 0.185, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority — [test comment as in outcome 4, analysis 3]; p = 0.164, ANCOVA

5. Secondary Outcome: Percent of Participants With WI-NRS 3-point Responder at Weeks 2, 4, and 10
Description: During the study, WI-NRS assessments were reported by the participant via eDiary once daily from screening/mid-screening visit through the follow-up visit. The Itch NRS is a validated, self reported, instrument for measurement of itch intensity and participants were asked to rate the intensity of their itch on an 11- point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity. A participant was a 3-point responder if their change from baseline is ≤ -3 (i.e. a decrease of at least 3).
Time Frame: At Weeks 2, 4, and 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Percentage of participants
  Percentage of responders at Week 2 | 8.11 | 11.89
  Percentage of responders at Week 4 | 18.24 | 20.03
  Percentage of responders at Week 10 | 25.65 | 37.58
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.283, Cochran-Mantel-Haenszel — P-value from a CMH test stratified by Baseline WI-NRS used for randomization stratification. Value has been adjusted for multiple imputation
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.701, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 10
Description: Dermatology Life Quality Index (DLQI) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the skin disease on a participant's QoL over the prior week. It is a ten item questionnaire that assesses overall QoL and six aspects that may affect QoL (symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment). The DLQI questions are rated by the participant as 0 (not at all) to 3 (very much). Scores range from 0 to 30 with higher scores indicating poor QoL.).
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Score on a scale | -4.4 (5.07) | -4.5 (5.14)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.797, ANCOVA — P-values, LS mean and SD from ANCOVA with treatment group and stratification factor as fixed effects, and baseline value as a covariate

7. Secondary Outcome: Change From Baseline in DLQI Question 1 to Week 10
Description: as for outcome 6
Time Frame: At Week 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Score on a scale | -0.6 (0.75) | -0.6 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.845, ANCOVA — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Change From Baseline in Investigator's Global Assessment of Prurigo Nodularis Stage (IGA PN-S) to Weeks 2, 4, and 10
Description: The IGA PN-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 (clear) to 4 (severe). Higher scores indicate severe prurigo nodularis.
Time Frame: At Weeks 2, 4 and 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Score on a scale
  Change from Baseline at Week 2 | -0.2 (0.43) | -0.2 (0.43)
  Change from Baseline at Week 4 | -0.4 (0.64) | -0.3 (0.64)
  Change from Baseline at Week 10 | -0.5 (0.77) | -0.5 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.385, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.786, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.502, ANCOVA — [p-value comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline in Investigator's Global Assessment of Prurigo Nodularis Activity (IGA PN-A) to Weeks 2, 4, and 10
Description: The IGA PN-A is an instrument used to assess the overall activity of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 (clear) to 4 (severe). Higher scores indicate severe prurigo nodularis.
Time Frame: At Weeks 2, 4, and 10
Population: Intent-to-Treat Population: included all randomized participants who were dispensed study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Score on a scale
  Change from Baseline at Week 2 | -0.2 (0.49) | -0.3 (0.49)
  Change from Baseline at Week 4 | -0.5 (0.68) | -0.5 (0.68)
  Change from Baseline at Week 10 | -0.7 (0.91) | -0.7 (0.92)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.197, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.694, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.916, ANCOVA — [p-value comment as in outcome 6, analysis 1]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. Severity of all AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03. During the period between informed consent and first study drug dose, only SAEs caused by a protocol-mandated intervention were collected.
Time Frame: From screening until the Follow-up (F/U) visit which occurred 35 days (+ 7 days) after the Week 10 visit or the last dose of study drug for participants who discontinued study drug early
Population: Safety population: included all treated participants with at least one post-baseline assessment or a reported TEAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 148 | 147
Participants
  Participants with any TEAE | 87 | 84
  Participants with any related TEAE | 24 | 30
  Participants with any serious TEAE | 2 | 5
  Participants with any related serious TEAE | 0 | 0
  Participants who Died | 0 | 0
  Participants who discontinued study drug | 4 | 13

ADVERSE EVENTS:
Time Frame: From screening until the Follow-up (F/U) visit which occurred 35 days (+ 7 days) after the Week 10 visit or the last dose of study drug for participants who discontinued study drug early.
Description: Adverse events (AEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. After informed consent was signed, but prior to initiation of study drug, only SAEs considered by the investigator to be caused by a protocol mandated intervention were collected.
Arm/Group | Placebo | Serlopitant 5 mg
All-Cause Mortality (participants affected / at risk) | 0/148 | 1/147
Serious Adverse Events (participants affected / at risk) | 2/148 | 5/147
Other Adverse Events (participants affected / at risk) | 33/148 | 31/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | Serlopitant 5 mg (N=147)
Coronary artery disease (Cardiac disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | Serlopitant 5 mg (N=147)
Fatigue (General disorders) | 6 | 7
Nasopharyngitis (Infections and infestations) | 22 | 15
Headache (Nervous system disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT03677401/Prot_001.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT03677401/SAP_000.pdf